CLINICAL TRIAL: NCT02950207
Title: Prospective Observational Study to Evaluate the Correlation Between Antitumor Activity of Hormone Therapy and the Expression of Micro-RNA (miRNA) 100
Brief Title: Prospective Observational Study of Antitumor Activity Correlation Between Hormonal Therapy and Expression miRNA100
Acronym: BC-P1-2013
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione del Piemonte per l'Oncologia (Other)
Responsible Party: Sponsor
Other Study IDs: BC-P1-2013
Record Dates: First submitted 2016-10-20; First posted 2016-11-01 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — MicroRNAs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: miRNA — miRNA extraction

SUMMARY:
Mono-centric, observational, prospective study, designed for pts with diagnosis of hormone-positive breast cancer to evaluate the correlation between the response to hormonal treatment indicated by the reduction of the level of Ki67 and miRNA100 in two groups of patients

DETAILED DESCRIPTION:
The potential role of miRNAs will be studied as a predictor of hormone sensitivity in hormone-positive breast carcinomas. The miRNA100 obtained on biopsy will be compared with the expression levels of those obtained from the surgically removed tumor, in order to assess the possible modulation of miRNA100 following hormonal treatment.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent
* Age greater than 18 years
* histological diagnosis of invasive carcinoma of the breast
* X-ray evidence (mammography and / or ultrasound) strongly suggestive for the presence of invasive breast cancer (BIRADS 4c or BIRADS 5) of greater than 15mm diameter.
* Carcinoma stage I (if diameter> 15 mm) or II, unresectable, or
* Carcinoma in stage II or III, operable as a result of presurgical therapy, or
* Carcinoma in IV debut stage, asymptomatic, with primary operable breast cancer, or as a result of presurgical therapy
* Positivity for the estrogen receptor and / or to the progestin defined as the expression of one or both hormone receptors in ≥10% of tumor cells
* Negativity for HER2
* Cell proliferation, defined as the percentage of Ki67 positive tumor cells,> 5% (corresponding to a value of 1.79 after log-normal transformation)
* Postmenopausal status
* Ability to take an oral therapy, in the absence of malabsorption syndrome known, previous stomach surgery or the small intestine
* Ability to perform the staging examinations and screening provided for in the
* Protocol
* Eastern Cooperative Oncology Group (ECOG) = 0
* The patients will have a normal bone marrow function, liver and kidney

Exclusion Criteria:

* Previous treatment for breast cancer with chemotherapy, lapatinib, trastuzumab, letrozole, anastrozole, exemestane or tamoxifen.
* Other cancers diagnosed in the last five years, with the exception of basal cell or squamous cell carcinoma of the skin, melanoma in situ or cervical cancer in situ.
* Premenopausal
* Known hypersensitivity to letrozole or to any of its excipients (for example: women with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or mal absorption of glucose / galactose).
* Evidence of a severe and poorly controlled systemic disease affecting the lung, heart, liver, kidney that may compromise adherence to treatment or an extended follow-up.
* Inflammatory bowel disease not controlled (eg Crohn's disease, ulcerative colitis).
* Active infection and / or inadequately controlled.
* Alteration of mental status, dementia, or any psychiatric condition that might impair the ability to consciously sign the informed consent.
* Breast cancer triple negative, or negative for both HER2 overexpression for the expression of hormone receptors.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: post menopausal hormone-positive breast cancer patients
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2014-01; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the efficacy | 42 months or until disease progression
  the natural logarithm value of Ki67 <1.0 defines the proliferative response to treatment. Response evaluation will be performed by measuring the reduction of Ki67 as a result of hormonal treatment according to a schedule defined on the basis of the stage of disease: patients with immediate operable cancer will be valued at the time of surgery (about 3 weeks).
  candidate patients to neoadjuvant hormone therapy and patients with stage 4 debut in hormonal therapy in advanced therapy (evaluation during the third week of starting treatment)

SECONDARY OUTCOMES:
Evaluation of Tolerability | 42 months or until disease progression
  The frequency and severity of adverse events will be evaluated based on the NCI-CTCAE v 4.0 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Filippo Montemurro, MD, Principal Investigator — FPO-IRCCS
Locations (1):
- Fondazione del Piemonte per l'Oncologia-IRCCS Candiolo, Candiolo, Turin, Italy

IPD SHARING:
Plan to Share IPD: No